CLINICAL TRIAL: NCT01786135
Title: A Phase 1, Open-Label, Dose-Escalation Study of SGN-CD19A in Patients With Relapsed or Refractory B-Lineage Non-Hodgkin Lymphoma
Brief Title: A Safety Study of SGN-CD19A for B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN19A-002
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-06

CONDITIONS: Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Precursor B-cell Lymphoblastic Leukemia-Lymphoma
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD19; B-Lineage Lymphoblastic Lymphoma; Burkitt Lymphoma; Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma; B-Cell Lymphoma; Drug Therapy; Monomethylauristatin F; Follicular Lymphoma Grade 3
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGN-CD19A (Experimental): SGN-CD19A (IV) once every 21 days (3 weeks) or 42 days (6 weeks)
  Interventions: Drug: SGN-CD19A

INTERVENTIONS:
Drug: SGN-CD19A — SGN-CD19A (IV) once every 21 days (3 weeks) or 42 days (6 weeks)

SUMMARY:
This is a phase 1, open-label, dose-escalation, multicenter study to evaluate the safety and tolerability of SGN-CD19A in patients with relapsed or refractory B-lineage non-Hodgkin lymphoma (B-NHL)

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of mantle cell lymphoma, follicular lymphoma Grade 3, diffuse large B-cell lymphoma (DLBCL), including transformed follicular histology, Burkitt lymphoma, or B-lineage lymphoblastic lymphoma
* Relapsed, refractory, or progressive disease following at least 1 prior systemic therapy. Patients with DLBCL or follicular lymphoma Grade 3 must have also received intensive salvage therapy.
* Eastern Cooperative Oncology Group status of 0 or 1
* Measurable disease

Exclusion Criteria:

* Allogeneic stem cell transplant (SCT)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month post last dose
Incidence of laboratory abnormalities | Through 1 month post last dose

SECONDARY OUTCOMES:
Objective response according to revised response criteria for malignant lymphoma (Cheson 2007) | Through up to approximately 6 week post last dose
Duration of response | Until disease progression or start of new anticancer treatment, an expected average of 6 months
Overall survival | Until death or study closure, an expected average of 1 year
Blood concentration of SGN-CD19A and metabolites | Through up to approximately 6 weeks post last dose
Incidence of antitherapeutic antibodies | Through up to approximately 6 weeks post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Ana Kostic, MD, Study Director — Seagen Inc.
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center / University of Texas, Houston, Texas